CLINICAL TRIAL: NCT01908985
Title: Ocular Fluorophotometry to Assess the Aqueous Humor Production for Patients With Glaucoma Treated With Cyclo-coagulation Using High Intensity Focused Ultrasound (HIFU).
Brief Title: Ocular Fluorophotometry for Glaucoma Treated With Cyclo-coagulation Using High Intensity Focused Ultrasound (HIFU).
Status: No longer available | Type: Expanded Access
Sponsor: EyeTechCare (Industry)
Responsible Party: Sponsor
Other Study IDs: EYEMUST-FLUO
Record Dates: First submitted 2013-07-24; First posted 2013-07-26 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2013-07

CONDITIONS: Refractory Open Angle Glaucoma
Keywords: glaucoma; high intensity focused ultrasound; aqueous humor; fluorophotometry
MeSH Terms: conditions — Glaucoma, Open-Angle; Glaucoma

INTERVENTIONS:
Procedure: high intensity focused ultrasound for cyclodestruction in the eye

SUMMARY:
Monocentric prospective study conducted in two phases evaluating the secretion and elimination of aqueous humor by fluorophotometry in patients with glaucoma treated with cyclo-coagulation with ultrasound.

Population selected:

- Patients with refractory open angle glaucoma despite previous treatments currently validated for glaucoma.

The purpose of our study is:

- To evaluate the mechanism of action of glaucoma treatment by cyclo-coagulation with high intensity focused ultrasound in studying the secretion and elimination of aqueous humor by fluorophotometry.

Planning:

* First phase: 2 patients (feasibility study) If reduction of at least 10% of the flow of aqueous humor production at one month in the first two patients in the feasibility study, further in second phase.
* Second phase: 6 patients

DETAILED DESCRIPTION:
Main outcome criteria:

Reduction of aqueous humor flow at 6 months compared with the pretreatment of aqueous humor flow.

ELIGIBILITY:
Inclusion Criteria:

* refractory primary open-angle glaucoma (POAG)
* IOP> 21 mm Hg and <32 mm Hg with an optimal treatment.
* Lack of history of cyclo-destruction of the ciliary body (laser diode, cold ...)
* Lack of intraocular surgery or laser therapy in the eye seen in the three months preceding the date of HIFU treatment.
* Male or female age (s) of at least 18 and able to give informed consent
* Patient who signed the informed consent form
* Patient affiliated to a social security scheme

Exclusion Criteria:

* History of glaucoma by placing a drainage implant (valves, pipes ...)
* previous refractive procedures preventing accurate measurement of intraocular pressure (PRK, LASIK)
* General treatment which may alter IOP began in the month before the HIFU procedure
* Patient monophthalmus
* thyroid orbitopathy
* History of ocular or retrobulbar tumor
* Cyclodialysis
* choroidal hematoma or uprising choroidal
* Anatomy of the eyeball inadequate treatment or medical device (eye too small or too large)
* Pregnancy, breastfeeding, lack of contraceptive use among women at risk of having a child
* Participation in another clinical investigation of a medical or surgical treatment can affect the intraocular pressure in the three months preceding the HIFU
* Patient minor or major protected by law

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult